CLINICAL TRIAL: NCT06371040
Title: Evaluate the Safety and Efficacy of CD19-BCMA Targeted CAR-T Therapy for Refractory, Generalized Myasthenia Gravis: A Single-center, Open-label, Single-arm, Dose-finding Study
Brief Title: Safety and Efficacy of CD19-BCMA Targeted CAR-T Therapy for Refractory Generalized Myasthenia Gravis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ting Chang, MD (Other)
Responsible Party: Sponsor-Investigator, Ting Chang, MD, Associate Professor, Tang-Du Hospital
Organization: Tang-Du Hospital (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: V1.0, CART-20230619
Record Dates: First submitted 2024-03-17; First posted 2024-04-17 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Myasthenia Gravis
Keywords: Generalized Myasthenia Gravis; CAR-T Therapy
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Intervention Model Description: CD19-BCMA Targeted CAR-T Dose 1 5.0 e5/ kg CD19-BCMA CAR-T positive T cells
  CD19-BCMA Targeted CAR-T Dose 2 1.5 e6/ kg CD19-BCMA CAR-T positive T cells
  CD19-BCMA Targeted CAR-T Dose 2 5 e6/ kg CD19-BCMA CAR-T positive T cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD19-BCMA Targeted CAR-T (Experimental)
  Interventions: Drug: CD19-BCMA Targeted CAR-T Dose 1; Drug: CD19-BCMA Targeted CAR-T Dose 2

INTERVENTIONS:
Drug: CD19-BCMA Targeted CAR-T Dose 1 — 5.0 e5/ kg CD19-BCMA CAR-T positive T cells
Drug: CD19-BCMA Targeted CAR-T Dose 2 — 1.5 e6/ kg CD19-BCMA CAR-T positive T cells
Drug: CD19-BCMA Targeted CAR-T Dose 2 — 5 e6/ kg CD19-BCMA CAR-T positive T cells

SUMMARY:
This study is a single-center, open-label, single-arm, dose-exploration study to evaluate the safety and preliminary effectiveness of CD19-BCMA CAR-T in the treatment of refractory, generalized myasthenia gravis. The study is a dose escalation trial in adult, refractory, systemic MG patients. The Keyboard method will be used to perform dose escalation to explore the maximum tolerated dose (MTD). A total of 12 MG patients who meet the inclusion criteria are expected to be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Study participants will be selected for this study only if they meet all of the following criteria:

  1. Age ≥18 years old and ≤80 years old;
  2. The subject signs the informed consent form, is willing and able to comply with the protocol, complete the research assessment and return for follow-up;
  3. To be diagnosed as a patient with systemic MG, the patient is required to have positive myasthenia-related antibodies (AChR-Ab, Musk-Ab or LRP4) on the basis of typical myasthenic symptoms;
  4. Evaluated by the researcher as refractory MG. Refractory MG is defined as:

     1. Treatment failed after receiving at least 2 immunosuppressants
     2. Definition of treatment failure: 1) Persistent weakness and impairment of daily activities; 2) MG aggravation and/or crisis during treatment; 3) Intolerance to immunotherapy due to side effects or comorbidities;
     3. Repeated plasma exchange (PE) or intravenous immune globulin (IVIg) treatment is required to control symptoms;
     4. The researchers believe that despite the current routine immunotherapy for patients, MG still imposes a large functional burden on patients.
  5. MGFA classification IIa~IVa at screening and baseline;
  6. QMGS score ≥11 points or MG-ADL score ≥5 points at screening and baseline, of which the eye score accounts for no more than 50%;
  7. Male study participants must agree to take contraceptive measures during the treatment period and within 1 year after receiving study treatment, and are prohibited from donating sperm throughout the study period;
  8. If you are a woman of childbearing potential (WOCBP), you must agree to take contraceptive measures during treatment and for at least 1 year after receiving study treatment. Participants must have a negative serum pregnancy test result during screening; a negative urine pregnancy test result must be confirmed before receiving CART for the first time.

Exclusion Criteria:

* Prior to screening and the baseline visit, study participants will not be eligible for inclusion in the study if they meet any of the following criteria:

  1. The researcher believes that there is any medical or mental condition that may harm the research participant or affect the research participant's ability to participate in this study; or any condition that the researcher believes is related to poor compliance;
  2. Women who are lactating or pregnant, or women who plan to become pregnant at any time within 12 months after receiving CART treatment, or who have a history of spontaneous abortion or induced abortion within 4 weeks before screening;
  3. Study participants have clinically relevant active infections (such as sepsis, pneumonia or abscess) or serious infections (resulting in hospitalization or requiring antibiotic treatment) within 4 weeks before screening;
  4. thymoma that underwent thymectomy within 6 months before baseline or was planned to undergo thymectomy during the study, or required chemotherapy and/or radiotherapy at any time;
  5. Investigator participants have received live attenuated vaccine vaccination within 8 weeks before screening; or plan to receive live vaccine vaccination within 8 weeks after treatment;
  6. Study participants have received rituximab treatment within 6 months before screening;
  7. Have received tocilizumab or eculizumab treatment within 3 months before screening;
  8. Have received intravenous human immunoglobulin, plasma exchange, or immunotherapy within 4 weeks before screening;
  9. Those with known serious underlying diseases, such as liver and kidney damage, blood diseases, previous severe cardiovascular disease, severe hypertension, diabetes, and poor blood pressure and blood sugar control;
  10. Unresected thymoma (Note: Subjects with benign thymoma resected more than one year before screening are eligible. Benign is defined as no known metastasis on pathological examination and no intracystic or extracystic Extension. Imaging studies must be performed during the screening period to assess thymic status).
  11. Any of the following laboratory abnormalities occur during the screening period (one repeat measurement can be performed during the screening period before randomization to confirm the results)

      1. Elevated liver enzymes (aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times the upper limit of normal (ULN)).
      2. Total bilirubin>1.5 times ULN
      3. Estimated glomerular filtration rate (eGFR) <45 mL/min/1.73 m2
      4. Abnormal PT or INR, or prolonged APTT >1.5 times ULN
      5. Neutrophil count <1000cell/ul
      6. Platelet count <50000/mm3
      7. Hemoglobin<8.0g/dl
  12. Those with a high-risk history of tuberculosis infection or acquired tuberculosis infection;
  13. Known immunodeficiency diseases, including human immunodeficiency virus (HIV) infection;
  14. Positive for hepatitis B surface antigen (HBsAg) during the screening period;
  15. Receive blood transfusion treatment 4 weeks before screening or during the screening period;
  16. Symptoms worsen rapidly during the lead-in period and enter crisis or pre-crisis state (MGFA IVb-V)
  17. Other circumstances in which the researcher deems it inappropriate to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Frequency, type, and severity of adverse events | From Baseline (Day 1) to Safety Follow-Up Visit (up to 4 weeks)
  Frequency, type, and severity of adverse events (according to the National Cancer Institute Common Terminology Criteria for Adverse Events CTCAE V5.0) occurring within 4 weeks after CD19-BCMA CAR-T infusion

SECONDARY OUTCOMES:
Frequency, type, and severity of abnormal laboratory indicators related to treatment | From Baseline (Day 1) up fo Follow-Up (up to 24 weeks)
  Frequency, type, and severity of abnormal laboratory indicators related to treatment (according to the National Cancer Institute Common Terminology Criteria for Adverse Events CTCAE V5.0)
Changes of blood pressure | From Baseline (Day 1) up fo Follow-Up (up to 24 weeks)
Changes of pulse rate | From Baseline (Day 1) up fo Follow-Up (up to 24 weeks)
Changes of weight | From Baseline (Day 1) up fo Follow-Up (up to 24 weeks)
Changes of Myasthenia Gravis Activities of Daily Living (MG-ADL) scores | From Baseline (Day 1) up fo Follow-Up (up to 24 weeks)
  Changes in MG-ADL scores [0-24 point] from baseline at 24 weeks after CD19-BCMA CAR-T infusion
Changes of Quantitative Myasthenia Gravis (QMG) scores | From Baseline (Day 1) up fo Follow-Up (up to 24 weeks)
  Changes in QMG scores [0-39 point] from baseline at 24 weeks after CD19-BCMA CAR-T infusion
Changes of Myasthenia Gravis Composite (MGC) scores | From Baseline (Day 1) up fo Follow-Up (up to 24 weeks)
  Changes in MGC scores [0-50 point] from baseline at 24 weeks after CD19-BCMA CAR-T infusion
Proportion of subjects who achieved improvement | From Baseline (Day 1) up fo Follow-Up (up to 24 weeks)
  Proportion of subjects who achieved improvement at 24 weeks after CD19-BCMA CAR-T infusion and sustained it for at least 4 weeks (clinical improvement difined as a ≥2-point reduction in the total MG-ADL score [0-24 point])
Time to achieve clinical improvement | From Baseline (Day 1) up fo Follow-Up (up to 24 weeks)
  Time to achieve clinical improvement (clinical improvement difined as a ≥2-point reduction in the total MG-ADL score [0-24 point])
Changes of myasthenia gravis-specific autoantibody titers | From Baseline (Day 1) up fo Follow-Up (up to 24 weeks)
  Changes from baseline in myasthenia gravis-specific autoantibody titers over 24 weeks after CD19-BCMA CAR-T infusion
Changes of immunoglobulins | From Baseline (Day 1) up fo Follow-Up (up to 24 weeks)
  Changes in immunoglobulins (IgG, IgM, IgA, IgE) within 24 weeks after CD19-BCMA CAR-T infusion

OTHER OUTCOMES:
Changes in proportion of peripheral blood immune cell | From Baseline (Day 1) up fo Follow-Up (up to 24 weeks)
  Changes in proportion of peripheral blood immune cell subsets of subjects after infusion of CD19-BCMA CAR-T
serum inflammatory markers levels | From Baseline (Day 1) up fo Follow-Up (up to 4 weeks)
  The levels of biomarkers used to evaluate safety and efficacy after infusion of CD19-BCMA CAR-T (ie, serum cytokine levels, serum inflammatory markers, plasma BCMA levels). Cytokines include at least IFNγ, IL-6, Soluble gp130, soluble IL-6R, TNFα, IL-2 and IL-10, other biomarkers and cytokines will be added based on the literature

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital, The Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Experimental data may be shared with the consent of the principal investigator
Supporting Information: CSR, Analytic Code
Time Frame: The entire study can be shared long-term after completion